CLINICAL TRIAL: NCT05092633
Title: Effect of Low Level Laser Therapy on Orthodontic Miniscrew Displacement
Acronym: Miniscrew
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Elzoheiry, Principal investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Effect of laser on mini screw
Record Dates: First submitted 2021-09-27; First posted 2021-10-25 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Orthodontic Appliance
Keywords: Miniscrew
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Will have miniscrew only without laser application
  Interventions: Device: Miniscrew
- Experimental (Experimental): Will have miniscrew and laser application
  Interventions: Device: Miniscrew

INTERVENTIONS:
Device: Miniscrew — Application of laser on miniscrew
  Other Names: Laser

SUMMARY:
EFFECT OF LOW LEVEL LASER THERAPY ON ORTHODONTIC MINISCREW DISPLACEMENT

DETAILED DESCRIPTION:
Miniscrews can achieve good anchorage for different types of tooth movements, as intrusion, retraction, and protraction. However, obtaining primary stability is a challenge in their clinical application.Low Level Laser Therapy is suggested to prevent miniscrew displacement. Also previous studies concluded that Low Level Laser Therapy has an effect in stabilizing miniscrew after direct application.

So the aim of this study is to assess the effect of Low Level Laser Therapy on displacement of miniscrews during canine retraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 22 years old.
* Permanent dentition.
* Class I Bimaxillary protrusion and class II devision 1 patients.
* Good oral hygiene.

Exclusion Criteria:

* Medically compromised patients.
* Chronic renal failure and hormonal disorders as thyroid and parathyroid.
* Regular use of steroids, barbiturates, anticonvulsants drugs, and thyroid hormone replacements.
* Tobacco smoking.
* Any disease or metabolic disorder that can affect bone physiology

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-09-26 (Actual); Primary Completion 2022-04-07 (Estimated); Study Completion 2022-05-05 (Estimated)

PRIMARY OUTCOMES:
effect of low level laser therapy on displacement of miniscrews | 4 months
  Miniscrews displacement will be assessed after four months of canine retraction using CBCT scan. The head and tail of miniscrew will be measured in relation to anterior nasal spine as a fixed reference point before and after retraction

SECONDARY OUTCOMES:
effect of LLL application on gingival condition around the miniscrew. | 4 months
  Gingival inflammation around miniscrew head will evaluated just after placement and at day 7 and 14 before application of retraction force and during days 21, 30, 60 which will be during the period of force application, based on modified gingival index with scores range from 0 to 3 as follows:Score 0 - no signs of inflammation (tissue around head is pink in color).
  Score 1 - mild inflammation (tissues are red in color, no bleeding sign). Score 2 - moderate inflammation (tissues are intense red in color, small bleeding signs).
  Score 3- severe inflammation (bleeding, evidence of swelling).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Elzoheiry, Study Director — Alexandria University
Locations (2):
- Egypt (2):
  - Alexandria University, Alexandria
  - AlexandriaU, Alexandria